CLINICAL TRIAL: NCT00866814
Title: A Prospective, Single Arm, Multi-Center Study Of Open Ventral Hernia Repair Utilizing The Bard Ventrio Hernia Patch
Brief Title: Study Of Hernia Repair Utilizing The Bard Ventrio Hernia Patch
Status: Completed | Type: Observational
Sponsor: C. R. Bard (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: DVL-HE004
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Results first posted 2012-05-21 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-10

CONDITIONS: Ventral Hernia
Keywords: hernia; open
MeSH Terms: conditions — Hernia, Ventral; Hernia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ventrio Group: Patients diagnosed with a ventral hernia requiring an open surgery for repair.
  Interventions: Device: Bard Ventrio Hernia Patch

INTERVENTIONS:
Device: Bard Ventrio Hernia Patch — The Ventrio Hernia Patch is a self-expanding, non-absorbable, sterile prosthesis for use in the reconstruction of soft tissue deficiencies, such as for the repair of hernias.

SUMMARY:
This study will collect data on patients undergoing hernia repair using the Bard Ventrio Hernia Patch. The study will evaluate hernia recurrence rates, operating time, quality of life and complications associated with the device and surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥ 18
2. Be able to undergo study procedures
3. Have signed an Informed Consent form (ICF)
4. Be diagnosed with a ventral hernia requiring an open surgery for repair.

Exclusion Criteria:

1. Patient is participating in another device or drug study.
2. Patient exhibits clinical symptoms indicating infected hernia site.
3. Patient currently has a clean contaminated or contaminated site.
4. Patient has a life expectancy less than 2 years at the time of enrollment.
5. Anything in the opinion of the Investigator that would preclude the use of the Ventrio Hernia Patch, or preclude the subject from completing the follow-up requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a diagnosis of ventral hernia will be screened for eligibility against the study protocol inclusion and exclusion criteria utilizing standard preoperative criteria (e.g. physical examination, blood work, medical evaluation, etc) which occurred within 30 days of the date of consent.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2009-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Iannitti, MD, FACS, Principal Investigator — Carolinas Medical Center
Locations (7):
- United States (7):
  - Sutter Medical Group GNS, Sacramento, California
  - Sacred Heart Health System, Inc., Pensacola, Florida
  - RUSH Univeristy Medical Center, Chicago, Illinois
  - Associated Surgical Group, Peoria, Illinois
  - Carolinas Medical Center, Charlotte, North Carolina
  - Gaston Memorial Hospital, Gastonia, North Carolina
  - Novant Clinical Research Institute, Winston-Salem, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From March 2009 through May 2010, a total of 119 patients were enrolled at 7 study centers in the United States.
Period: Overall Study
Arm/Group | Ventrio Group
Started | 119
Completed | 99
Not Completed | 20
Not completed — Lost to Follow-up | 12
Not completed — Adverse Event | 2
Not completed — Physician Decision | 1
Not completed — Death | 1
Not completed — No longer wished to participate | 1
Not completed — Unable to meet follow-up requirements | 2
Not completed — Moved to area without study site | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ventrio Group
Number analyzed (Participants) | 119
Age Continuous [Mean (Standard Deviation); unit: years] | 55.8 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 48
Region of Enrollment [Number; unit: participants]
  United States | 119
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 33.5 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint is the Rate of Hernia Recurrence in Study Patients.
Description: A recurrent hernia is a hernia, confirmed by the investigator at any point within the first year after surgery, in the same location as the hernia repaired in the index procedure.
Time Frame: 1 year post surgery
Population: All enrolled patients.
Measure: Number; unit: participants
Arm/Group | Ventrio Group
Number analyzed (Participants) | 119
participants | 0

2. Secondary Outcome: Perioperative Complications Will be Assessed by Evaluation of the Procedural and Device Related Adverse Events (AEs) Collected From the Time Surgery is Initiated Until the Day the Patient is Discharged From the Hospital.
Description: In this study, a complication was defined as any adverse event that was assessed by the Investigator as either possibly or definitely related to the study procedure or the study device.
Time Frame: From the time of surgery to hospital discharge, an average of 1-2 days
Population: All enrolled patients.
Measure: Number; unit: Complication events
Arm/Group | Ventrio Group
Number analyzed (Participants) | 119
Complication events | 4

3. Secondary Outcome: Short-term Complications Will be Assessed by Evaluation of the Procedural and Device Related AEs Collected From the Day After the Patient is Discharged From the Hospital Until 21 Days Post Procedure.
Description: as for outcome 2
Time Frame: Hospital discharge through 21 days post surgery
Population: All enrolled patients.
Measure: Number; unit: Complication events
Arm/Group | Ventrio Group
Number analyzed (Participants) | 119
Complication events | 10

4. Secondary Outcome: Long-term Complications Will be Assessed by Evaluation of the Procedural and Device Related AEs Collected After 21 Days up to 1 Year.
Description: as for outcome 2
Time Frame: 22 days post surgery through 1 year post surgery
Population: All enrolled patients.
Measure: Number; unit: Complication events
Arm/Group | Ventrio Group
Number analyzed (Participants) | 119
Complication events | 6

5. Secondary Outcome: Quality of Life Will be Assessed at Baseline Through 1 Year Utilizing the Carolinas Comfort Scale Survey
Description: Mean Quality of Life scores at each study visit for the "sensation of mesh," "pain," and "movement limitation" components of the Carolinas Comfort Scale are reported. Patient responses are provided on a ordinal scale from 0-5 indicating increasing severity of symptoms with 0 representing no symptoms and 5 representing disabling symptoms. Sensation of mesh was not evaluable at baseline and therefore, scores are reported starting at 2 weeks post study procedure.
Time Frame: Baseline and post-surgery at week 2, month 6 and month 12
Population: All enrolled patients with QOL scores at each visit.
Measure: Mean (Standard Deviation); unit: units on a scale (0-5)
Arm/Group | Ventrio Group
Number analyzed (Participants) | 119
units on a scale (0-5)
  Sensation of mesh: week 2 | 0.7 (1.2)
  Sensation of mesh: month 6 | 0.3 (0.7)
  Sensation of mesh: month 12 | 0.1 (0.5)
  Pain: baseline | 1.3 (1.3)
  Pain: week 2 | 1.6 (1.4)
  Pain: month 6 | 0.3 (0.6)
  Pain month 12 | 0.2 (0.6)
  Movement limitations: baseline | 1.1 (1.3)
  Movement limitations: week 2 | 1.4 (1.4)
  Movement limitations: month 6 | 0.2 (0.6)
  Movement limitation month 12 | 0.1 (0.5)

6. Secondary Outcome: Procedure Time
Description: Procedure time will be defined as beginning when the investigator makes the initial incision and ending when the skin closure is completed.
Time Frame: Day of surgery
Population: All enrolled patients.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ventrio Group
Number analyzed (Participants) | 119
minutes | 42.8 (19.8)

ADVERSE EVENTS:
Time Frame: Protocol defined adverse events were collected beginning at the time of the study repair procedure (first incision) through study completion or withdrawal.
Description: Adverse events were defined as any undesirable clinical event occurring in the abdominal wall or involving abdominal organs and/or judged to be related to the surgical procedure or Ventrio hernia patch.
Arm/Group | Ventrio Group
Serious Adverse Events (participants affected / at risk) | 8/119
Other Adverse Events (participants affected / at risk) | 14/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ventrio Group (N=119)
Consitpation (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) — Subject's study device removed as a result of postoperative wound infection and seroma.
Wound infection (Infections and infestations) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) — Subject's study device removed as a result of postoperative wound infection and seroma.
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Bile duct cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) — Study device was removed approximately 6 months post procedure as a result of procedural pain.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ventrio Group (N=119)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Application site vesicles (General disorders) | 1 (1)
Hernia (General disorders) | 1 (1) — Patient developed a new (non-study) hernia at a different surgical site as the result of a non-study procedure.
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) — Two adverse events were identified by clinical monitoring but not reported in the clinical database by the study site (one event of postoperative ileus and one event of abdominal pain).
Seroma (Injury, poisoning and procedural complications) | 5 (5)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was designed as a single arm observational trial without predefined statistical hypotheses (theories) to test; therefore, data can only be described and no treatment comparisons or conclusions can be made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days